CLINICAL TRIAL: NCT04444999
Title: Carbon Dioxide Guided Angiography in Endovascular Abdominal Aortic Aneurysm Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD.19.11.248 - 2019/11/01
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: carbon dioxide (CO2) digital subtraction angiography (DSA) to guide endovascular aneurysm repair (EVAR(
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular abdominal aortic aneurysm repair (Experimental): a type of endovascular surgery used to treat pathology of the aorta, most commonly an abdominal aortic aneurysm (AAA).
  Interventions: Procedure: Carbon Dioxide Angiography

INTERVENTIONS:
Procedure: Carbon Dioxide Angiography — • Automated carbon dioxide angiography: Patients are placed in the Trendelenburg position with the feet elevated of 10 º degrees. Carbon Dioxide automatic injection will be performed by digital Angiodroid injection system

SUMMARY:
Endovascular aneurysm repair (EVAR) has lower short-term morbidity and mortality than open surgery. Intra-arterial contrast agents are an important component of successful EVAR as the tool of choice for preoperative evaluation of aortic aneurysm morphology as well as precise sizing and intraoperative visualization of the ostia of the renal and hypogastric arteries for graft replacement. Although iodinated contrast (IC) is overwhelmingly the most common contrast agent, the perioperative use of IC agents is not recommended in patients with renal dysfunction or allergies to IC The aim of this study was to evaluate feasibility, efficacy and safety of carbon dioxide (CO2) digital subtraction angiography (DSA) to guide endovascular aneurysm repair (EVAR) in a cohort of patients with abdominal aortic aneurysm

DETAILED DESCRIPTION:
INTRODUCTION:

Endovascular aneurysm repair (EVAR) has lower short-term morbidity and mortality than open surgery. Intra-arterial contrast agents are an important component of successful EVAR as the tool of choice for preoperative evaluation of aortic aneurysm morphology as well as precise sizing and intraoperative visualization of the ostia of the renal and hypogastric arteries for graft replacement. Although iodinated contrast (IC) is overwhelmingly the most common contrast agent, the perioperative use of IC agents is not recommended in patients with renal dysfunction or allergies to IC.

Many strategies have been proposed with the aim of reducing IC developed, such as the use of intravascular ultrasound, high-quality 3-dimensional imaging techniques, and fusion of preoperative and intraoperative imaging. However, despite reports of various methods of renal protection, including the use of perioperative hydration, acetylcysteine, mannitol, dopamine, and fenoldopam, the effects of these methods are controversial.

Carbon dioxide (CO2)-guided angiography is an alternative contrast approach first described for diagnostic purposes by Hawkins. Although many studies have demonstrated the safety and effectiveness of CO2-EVAR and its noninferiority to Iodinated Contrast Angiography during EVAR.

Intravascular ultrasound (IVUS) has been used as an alternative to IACA(intra-arterial contrast agents). Originally, IVUS images had low accuracy, but recent improvements have resulted in very high-quality images of intra-aortic structures, which makes the use of IACA(intra-arterial contrast agents) almost unnecessary. An additional advantage of IVUS is that it facilitates the precise placement of stent grafts, because it is more accurate in locating hypogastric arteries and renal arteries which have parallax from the anteroposterior (A-P) view rather than from angiography. In this study, investigators will compare Carbon Dioxide Guided Angiography in relation to Iodinated Contrast Angiography during EVAR.

Aim of the work The aim of this study was to evaluate feasibility, efficacy and safety of carbon dioxide (CO2) digital subtraction angiography (DSA) to guide endovascular aneurysm repair (EVAR) in a cohort of patients with abdominal aortic aneurysm.

Outcome Primary outcomes: Validity of CO2 in Visualizing of Renal and hypogastric arteries. Neck of the aneurysm measurements. Endoleaks Secondary outcomes: Safety of CO2

Patients and methods Study location: The study will be conducted at the department of vascular surgery in Mansoura university hospitals Study population: The study will be conducted in patients with Abdominal Aortic Aneurysm.

Type of the study: Evaluation of diagnostic imaging. Duration of therapy: Two year 2019-2021. Sample size: It will include all patients presented to our department fulfilling the inclusion criteria; sample size will be 50 patients.

n=(Z^2 p(1-p))/d^2 Where: Z= 1.96 at 95% confidence level, P= expected prevalence, d= precision (margin of error) Inclusion criteria Age 18 years old. Less than 50 years old Abdominal Aortic above Aneurysm candidate for EVAR. Exclusion criteria: previous abdominal aortic surgery, , mycotic aneurysm and secondary intervention.

Data collection: The demographics, Symptoms and preoperative clinical data will be collected Consent: Patients after signing informed consent that possible complication from the procedure ought to happen and what are the alternatives.

Technique:

All procedures are performed using two angiographic methods in each procedure: automated conventional ICM digital subtraction angiography (DSA) and CO2 automated DSA, in a Philips hybrid operating theatre. IVUS method (instead of ICM) will be used in chronc kidney disease patients Proximal and distal sealing zone are evaluated before and after endograft deployment, for diagnostic and completion evaluation respectively, by both imaging methods.

The presence of endoleaks will be also evaluated at the completion angiography, by both methods.

The angiographic results that will be obtained by CO2 and ICM will be compared. Preoperative imaging will be performed by contrast enhanced computed tomography (CTA); analyzed with dedicated software for vessels analysis. centerline will be manually calculated by selecting points at the center of aorta and iliac arteries using multi planar reconstructions (axial, sagittal and coronal views).

Abdominal aortic aneurysm volumetric evaluation is performed by selecting points of the external aortic wall (AAA total volume) and of the internal aortic lumen (AAA true luminal volume) from the lower renal artery to the aortic bifurcation, using a dedicated software of volumetric CTA analysis (3MensioTM).

Conventional contrast media angiography: Iodinate contrast media DSA will be performed by automatic and manual injection. For the automatic DSA, isotonic ICM is injected trough a pigtail catheter (5F/65 mm length) positioned just above the renal arteries, using automated injector. During each procedure two automated ICM DSA, with a volume of 20 mL at a rate of 14 mL/s, are performed: a diagnostic injection before the deployment of the endograft, in order to visualize the proximal sealing zone, the aortic bifurcation and the distal sealing zone, and a completion angiography to confirm the technical success and to evaluate the presence of endoleaks. Manual retrograde injections (3 mL ICM each) are performed from the femoral access by 10 F /11mm length sheet to visualize the hypogastric arteries origin and confirm the distal sealing zone just before the limb deployment.

Intravascular ultrasound (IVUS) will have been used as an alternative to iodinated contrast in if the iodinated contrast contraindicated patients. The IVUS procedure steps used are summarized here.

First, the bilateral common femoral arteries were exposed and a 9-F sheath introducer the lowest profile adjusted to the 8.2-F of the outer diameter of the IVUS transducer is inserted retrograde. A soft guidewire is used to introduce a calibrated pigtail catheter, graduated in centimetres, up to the thoracic aortic arch. The guidewire is then replaced with a stiff wire followed by IVUS insertion. IVUS is used to locate the renal arteries and hypogastric arteries by mapping them on the monitor; then, IVUS is switched to the calibrated catheter to determine the length of the main body.

IVUS is introduced using the monorail system. After deployment of the main body, the soft guidewire is cannulated into the contralateral limb. The guidewire is replaced with the stiff wire, followed by the IVUS insertion. The length of the contralateral site is determined by measuring the length from the edge of the main body to the site of the hypogastric ostium. Using the same technique, investigators will estimate the stent graft length with the calibrated catheter. Automated carbon dioxide angiography: Patients are placed in the Trendelenburg position with the feet elevated of 10 º degrees. Carbon Dioxide automatic injection will be performed by digital Angiodroid injection system (Angiodroid SRL, San Lazzaro, Bologna, Italy) connected to the sidearm of 10F/11mm length sheet. Ten milliliters of CO2 are infused to fill the tubing with gas and eliminate the air. Then by apposite manipulation of the stopcocks, the sheath is back-bled through its sidearm, and CO2 infused, creating a blood-CO2 interface with no air in the system 12. The 10F sheet is positioned at the level of the external iliac artery at the contralateral access of the main body. Each injection volume will be 100 mL of CO2 and the injection pressure is 300 mmHg (Figure 1D). To avoid gas fragmentation, the catheter will be purged prior to each injection and delivery is in a continuous controlled fashion. During each procedure a diagnostic evaluation, before the deployment of the endograft, an angiography to visualize the hypogastric arteries origin and a completion angiography, is performed after the positioning of the endograft. Both the endograft deployment angiography and the completion angiography will be performed maintaining a constant blood systolic pressure, between 100 and 120 mmHg.

Operative technique: All the procedures are performed in a Philips hybrid operating theatre and all angiograms are obtained using the Integris Allura 12 DSA. Bilateral common femoral artery access is obtained through surgical cut down under spinal or general anesthesia. According with the vertebral bone landmarks, identified pre-operatively, the main-body endograft is advanced up to the juxta-renal aortic segment. An angiographic evaluation is performed before the endograft deployment. After contra-lateral gate cannulation, a marked pig tail will be used to measure the iliac limb length and to identify the origin of the hypogastric artery from the contralateral access. When a trimodular endograft is deployed, the same maneuver will be performed for the ipsilateral access. Patients considered at high risk for persistent type II endoleak (ELII) underwent intraoperative AAA sac embolization as reported in a previous experience. After the endograft deployment a completion angiography is performed in all cases.

Endpoints and definition Primary endpoints are to determine the efficacy of CO2 automated DSA in proximal/distal sealing zone evaluation and endoleaks detection, in comparison with ICM.

Secondary endpoint is to evaluate the safety of CO2 standardized automated injection (any side effects).

Patients are defined fit for standard EVAR when proximal and distal neck length was ≥ 15 mm and aortic neck β angle and angles at the level of iliac arteries were < 60°.

Diagnostic angiography is defined as the first angiography performed with the main body advanced at the level of the lower renal artery according to bone landmarks, just before its deployment, in order to visualize the optimal proximal sealing zone.

The intraoperative proximal sealing zone evaluation is defined effective when the lower renal artery and the proximal aortic neck just below it, are correctly visualized.

The intraoperative distal sealing zone evaluation is defined effective if the origin of the hypogastric artery and the distal segment of the common iliac artery just above it, are visualized.

Technical success (TS) is defined as the complete endograft deployment with patency of renal and hypogastric arteries, absence of type I/III endoleaks and iliac leg kinking or stenosis, no conversion to OR or 24-hour mortality. Endoleaks are defined according to White and May classification .

CO2 side effects (CO2 narcosis) are defined as any adverse events correlate to CO2 automated injection. As reported in literature, abdominal pain, transient hypotension, nausea, ischemic colitis occurring intraoperatively or within 30 minutes from the procedure, are considered adverse events correlate to CO2.

Follow up Every patient will be followed first week and month, then every 3 months For at least 6 months.

Evaluation made by CTA or duplex ultrasonography

Statistical analysis:

The clinical characteristics of the study population is summarized by descriptive statistics. The following tests Fisher's exact test and the Mann-Whitney U test; used for categorical and continuous variables, respectively. Sensitivity and specificity will measures of the performance of the test Individual differences were considered to be statistically significant at p < 0.05 Continuous data are presented as median and interquartile range (IQR).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old. Abdominal Aortic above Aneurysm candidate for EVAR

Exclusion Criteria:

* previous abdominal aortic surgery, , mycotic aneurysm and secondary intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Validity of Carbon Dioxide angiography in Visualizing of Renal and hypogastric arteries. | 6 months
  Visualizing of Renal and hypogastric arteries.
Validity of Carbon Dioxide angiography in Visualizing Neck of the aneurysm measurements. | 6 months
  measuring the supra renal and infra renal neck measurements
Validity of Carbon Dioxide angiography in Visualizing Endoleaks | 6 months
  Endoleaks occur when blood leaks back into an aneurysm sac following an endovascular aneurysm repair (EVAR) procedure-one of the procedure's most common complications.

SECONDARY OUTCOMES:
Safety of Carbon Dioxide angiography at Endovascular aortic aneurysm repair | 6 months
  Adverse effects of Carbon Dioxide angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura, Al Mansurah, Mansoura University, Egypt

IPD SHARING:
Plan to Share IPD: No